CLINICAL TRIAL: NCT05873244
Title: Epigenetic Therapeutics to Overcome Resistance Against Immune Checkpoint Inhibitors in Hepatocellular Carcinoma: A Proof-of-concept Clinical Trial
Brief Title: CXD101 in Immunotherapy-related Liver Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephen Chan Lam (Other)
Responsible Party: Sponsor-Investigator, Stephen Chan Lam, Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC074
Record Dates: First submitted 2023-05-03; First posted 2023-05-24 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: HCC
MeSH Terms: interventions — lenvatinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment arm (Experimental): * Zabadinostat (CXD101) at 20mg twice daily per orally Day 1-5 every 3 weeks
  * Geptanolimab at 3mg/kg given intravenously every 2 weeks
  Interventions: Drug: Zabadinostat (CXD101) and Geptanolimab
- Control arm (Other): Clinicians' choice of TKI at corresponding recommended dosage:
  * Lenvatinib at 8mg daily for patients with body weight <60kg or 12mg daily with body weight ≥ 60kg
  * Sorafenib at 400mg twice daily
  Interventions: Drug: Lenvatinib and Sorafenib

INTERVENTIONS:
Drug: Zabadinostat (CXD101) and Geptanolimab — * Zabadinostat (CXD101) at 20mg twice daily per orally Day 1-5 every 3 weeks
  * Geptanolimab at 3mg/kg given intravenously every 2 weeks
  Arms: Experiment arm
Drug: Lenvatinib and Sorafenib — Clinicians' choice of TKI at corresponding recommended dosage:
  * Lenvatinib at 8mg daily for patients with body weight <60kg or 12mg daily with body weight ≥ 60kg
  * Sorafenib at 400mg twice daily
  Arms: Control arm

SUMMARY:
For hepatocellular carcinoma (HCC), durable responses and improved survivals have been reported in clinical trials on immune checkpoint inhibitor (ICI)-based treatment. However, resistance to ICI is increasingly encountered in clinical practice in HCC patients.

Various approaches are currently evaluated in clinical setting to tackle acquired resistance during treatment of ICIs in HCC.

Our group has a track record of studying the role of histone deacetylases (HDACs) in mediating resistance to ICI in HCC. First, based on single-cell sequencing data of serial biopsy of tumor in our phase II clinical trial on pembrolizumab in HCC (NCT03419481), the investigators reveal an upregulation of class 1 HDAC in patients with acquired resistance to pembrolizumab, which was associated with reduced lymphoid/myeloid cellular ratio in the tumor. Further, the investigators showed that HDAC8, a class 1 HDAC, could diminish the efficacy of anti-programmed cell death (ligand)-1 (PD[L]-1) by the mechanism of T-cell exclusion from the tumor environment (SciTranl Med. 2021;13:online). Finally, the investigators combine CXD101, a potent selective class I HDAC inhibitor, with anti-PD(L)-1 in orthotopic immunocompetent HCC mouse model with resistance to anti-PD(L)-1 treatment and find that the combination regimen could reverse the resistance phenotype and significantly improve survivals of mice than either CXD101 or anti-PD(L)-1 alone.

DETAILED DESCRIPTION:
To move from bench to clinic, it is crucial to validate the above in HCC patients demonstrating resistance to ICI-based treatment. In this grant, the investigators propose a randomized phase II clinical trial in patients with HCC who developed progressive disease to prior regimen containing anti-PD(L)-1. The investigators have already secured support of study medications from two pharmaceuticals to provide class 1 HDAC inhibitor and anti-PD1, respectively. Patients were randomized 1:1 to two study arms: the experiment arm consists of CXD101 20mg twice daily Day 1-5 every 3 weeks and an anti-PD1, geptanolimab at 3mg/kg Day 1 every 2 weeks. The dose of CXD101 has already been confirmed to be safe to combine with anti-PD1 in phase I/II studies in cancer patients. The control arm consists of investigators' choice of lenvatinib or sorafenib which are both considered standard treatment after failure with first-line atezolizumab-bevacizumab or other anti-PD(L)-1-based treatment. The primary endpoint is progress-free survival. Along the clinical trial, tumor biopsy will also be conducted at baseline and 6-week post-treatment to explore potential predictive biomarkers. Results of the study not only act as proof-of-concept but also potentially develop a novel treatment combination to tackle resistance to anti-PD(L)-1 treatment in HCC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HCC according to the AASLD guideline20
* Prior treatment with systemic treatment consisting of immune checkpoint inhibitors (anti-PD1, anti-PDL1 or anti-CTLA4)
* The duration of previous ICI must be 6 weeks or longer to avoid chance of pseudo-progression
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-1
* Adequate hematological function:
* Absolute neutrophil count (ANC) ≥ 1.5 x109/L; Platelets ≥ 100 x 109/L and Hemoglobin ≥ 8g/dL
* Adequate renal function:
* Urine protein/creatinine ratio ≤ 1 mg/mg (≤ 113.1 mg/mmol) or 24-hour urine protein < 1g
* Serum creatinine ≤ 1.5 × upper limit of normal or calculated creatinine clearance ≥ 40 mL/min (according to the Cockcroft-Gault equation)
* Adequate hepatic function parameters:
* Total bilirubin ≤ 2 mg/dL (≤ 34.2 μmol/L)
* Serum albumin ≥ 2.8 g/dL (≥ 28 g/L)
* Alanine aminotransferase (ALT) < 3.0 upper limit of normal (ULN)

Exclusion Criteria:

* Previous development of severe autoimmune complications from immune checkpoint inhibitors
* History of moderate to sever autoimmune disease requiring steroid use
* History of organ transplant
* Prior use of lenvatinib or sorafenib
* Disease involvement/thrombosis of major vessels (including main trunk of portal vein, inferior vena cava or pulmonary artery)
* More than two lines of systemic therapy (i.e., study treatment must be second-line or third-line treatment)
* Clinically significant bleeding events (eg.. esophageal varices) within 3 months
* Moderate or severe ascites
* Child-pugh B or C hepatic function
* Systolic blood pressure of 200mmHg or higher
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The progression-free survival in HCC patients treated with CXD101 plus Geptanolimab and control arm | 2 years

SECONDARY OUTCOMES:
The overall survival in HCC patients treated with CXD101 plus Geptanolimab and control arm | 2 years
The radiological response rate in HCC patients treated with CXD101 plus Geptanolimab and control arm | 2 years
The time-to-progression in HCC patients treated with CXD101 plus Geptanolimab and control arm | 2 years
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong
  - School of Biomedical Science, The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tu Y, Wu H, Zhong C, Liu Y, Xiong Z, Chen S, Wang J, Wong PP, Yang W, Liang Z, Lu J, Chen S, Zhang L, Feng Y, Si-Tou WW, Yin B, Lin Y, Liang J, Liang L, Vong JSL, Ren W, Kwong TT, Leung H, To KF, Ma S, Tong M, Sun H, Xia Q, Zhou J, Kerr D, La Thangue N, Sung JJY, Chan SL, Cheng AS. Pharmacological activation of STAT1-GSDME pyroptotic circuitry reinforces epigenetic immunotherapy for hepatocellular carcinoma. Gut. 2025 Mar 6;74(4):613-627. doi: 10.1136/gutjnl-2024-332281. PMID 39486886